CLINICAL TRIAL: NCT03068143
Title: A Muti-centre Prospective Observational Study on Postoperative Temperature Monitoring In Patients With Brain Trauma
Brief Title: Postoperative Temperature Monitoring In Brain Trauma
Acronym: PTMIBT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BT-201607
Record Dates: First submitted 2017-02-21; First posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Brain Injuries, Traumatic; Body Temperature Changes
MeSH Terms: conditions — Brain Injuries, Traumatic; Body Temperature Changes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study is designed to investigate the relationship between brain temperature, axillary temperature, rectal temperature, and bladder temperature of postoperative patients with brain trauma, and the relationship between brain temperature and prognosis. This study is conducted based on the following important assumptions. First, brain temperature of postoperative patients with brain trauma should be higher than the axillary temperature, rectal temperature and bladder temperature. Second, the consistency of brain temperature and bladder temperature is better than the consistency of brain temperature and axillary temperature, as well as that of brain temperature and rectal temperature. Third, brain temperature can help clinicians to predict the prognosis of patients with brain trauma. Therefore, brain temperature monitoring is significant in postoperative intensive care and treatment of patients with brain trauma.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or radiological diagnosis is brain trauma;
* The patient has surgical indications, and the patient or his/her family are willing to undergo operation including brain temperature monitoring probe implantation;
* Informed consent is obtained from the patient's family.

Exclusion Criteria:

* At the time of admission there are serious systemic diseases, including severe infections, immune system diseases, blood system diseases, infectious diseases, severe liver and kidney dysfunction, malignant tumors, etc;
* Pregnant or lactating women;
* There are other brain tumors or cerebrovascular disease in the brain at the same time;
* There is a history of drug or alcohol abuse;
* Within 3 months before admission, live vaccines were inoculated.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients with brain trauma
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Change of Brain Temperature | Change from Baseline Brain Temperature at 1 week
Change of Axillary Temperature | Change from Baseline Axillary Temperature at 1 week
Change of Rectal Temperature | Change from Baseline Rectal Temperature at 1 week
Change of Bladder Temperature | Change from Baseline Bladder Temperature at 1 week
Glasgow Outcome Scale | 1 month
  An objective assessment of the recovery of patients with brain trauma

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Hayward JN, Baker MA. A comparative study of the role of the cerebral arterial blood in the regulation of brain temperature in five mammals. Brain Res. 1969 Dec;16(2):417-40. doi: 10.1016/0006-8993(69)90236-4. No abstract available. PMID 4311724
- [Background] Mellergard P, Nordstrom CH. Intracerebral temperature in neurosurgical patients. Neurosurgery. 1991 May;28(5):709-13. PMID 1876249
- [Background] Mellergard P, Nordstrom CH, Messeter K. Human brain temperature during anesthesia for intracranial operations. J Neurosurg Anesthesiol. 1992 Apr;4(2):85-91. doi: 10.1097/00008506-199204000-00003. PMID 15815447
- [Background] Hirashima Y, Takaba M, Endo S, Hayashi N, Yamashita K, Takaku A. Intracerebral temperature in patients with hydrocephalus of varying aetiology. J Neurol Neurosurg Psychiatry. 1998 Jun;64(6):792-4. doi: 10.1136/jnnp.64.6.792. PMID 9647313
- [Background] Camboni D, Philipp A, Schebesch KM, Schmid C. Accuracy of core temperature measurement in deep hypothermic circulatory arrest. Interact Cardiovasc Thorac Surg. 2008 Oct;7(5):922-4. doi: 10.1510/icvts.2008.181974. Epub 2008 Jul 25. PMID 18658167
- [Background] Henker RA, Brown SD, Marion DW. Comparison of brain temperature with bladder and rectal temperatures in adults with severe head injury. Neurosurgery. 1998 May;42(5):1071-5. doi: 10.1097/00006123-199805000-00071. PMID 9588552
- [Derived] Weng WJ, Yang C, Huang XJ, Zhang YM, Liu JF, Yao JM, Zhang ZH, Wu XS, Mei T, Zhang CD, Jia J, Shi XF, Mao Q, Feng JF, Gao GY, Jiang JY. Effects of Brain Temperature on the Outcome of Patients with Traumatic Brain Injury: A Prospective Observational Study. J Neurotrauma. 2019 Apr 1;36(7):1168-1174. doi: 10.1089/neu.2018.5881. Epub 2018 Oct 10. PMID 30215286